CLINICAL TRIAL: NCT04818801
Title: A Phase 1, First-in-human, Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of ReCOV, a Vaccine for COVID-19, in Healthy Adult Subjects
Brief Title: Safety, Reactogenicity and Immunogenicity Study of ReCOV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jiangsu Rec-Biotechnology Co., Ltd. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT61101
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant two-component COVID-19 vaccine (CHO cell) (Experimental): Participants received Recombinant two-component COVID-19 vaccine (CHO cell) 0.5ml reconstituted by adjuvant solution, 2 shots at a interval 21 days, intramuscular injection
  Interventions: Biological: Recombinant two-component COVID-19 vaccine (CHO cell)
- Placebo (Placebo Comparator): Participants received placebo of 0.5ml normal saline (0.9% sodium chloride solution), 2 shots at a interval 21 days, intramuscular injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Recombinant two-component COVID-19 vaccine (CHO cell) — The spike (S) protein is the main surface antigen of SARS-CoV-2, mediates entry of SARS CoV-2 into cells expressing the angiotensin-converting enzyme 2 (ACE2). The RBD interacts with ACE2 and can generate potent neutralizing anti-RBD antibodies.
  Other Names: ReCOV
  Arms: Recombinant two-component COVID-19 vaccine (CHO cell)
Other: Placebo — Normal saline (0.9% sodium chloride solution),
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the pathogen that causes a coronavirus-associated acute respiratory disease called coronavirus disease 19 (COVID-19), which is spreading all over the world. This virus can cause acute respiratory distress syndrome (ARDS) with a high fatality rate.

In this phase I first-in-human clinical trial, healthy volunteers in two different age cohorts and two dose cohorts will be vaccinated twice with the candidate vaccine ReCOV.

The aim of the study is to assess the safety and reactogenicity of the candidate vaccine and to characterize its immunogenicity.

DETAILED DESCRIPTION:
A total of 100 participants will receive the following vaccine regime:

First, 20 young adult participants (18 to 55 years old) will receive 20μg of ReCOV vaccine on days 0 and 21.

Then, 20 young adult participants (18 to 55 years old) will receive 40μg of ReCOV vaccine on days 0 and 21, and 20 old adult participants (56 to 80 years old) will receive 20μg of ReCOV vaccine on days 0 and 21.

Finally, 20 old adult participants (56 to 80 years old) will receive 40μg of ReCOV vaccine on days 0 and 21.

In the same time, 8 participants for each cohort, total 32 participants will receive 0.5ml of normal saline on days 0 and 21.

Safety and immunogenicity data will be collected throughout the study, which concludes at 12 month after the second dose.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if ALL of the following criteria apply at any time starting from Screening up to Day 1 prior to IP administration:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol.
2. Male or female subjects who are ≥18 years old at the time of Screening (signing the ICF):

   1. For the younger adult group: 18 to 55 years, inclusive
   2. For the older adult group: ≥56 to <80 years
3. Have a body mass index (BMI) between 18.5 and 35.0 kg/m2.
4. Subjects who are of general good health according to the Investigator's assessment, based on a complete medical history without major pathology, and as determined by medical evaluation (including physical examination, electrocardiogram (ECG), vital signs, and clinical laboratory tests). Subjects in the older adult population who have medically stable, well-controlled comorbidities may be enrolled at the discretion of the Investigator.

   NOTE: All clinical laboratory values should be within reference ranges unless confirmed by Investigator or delegate as not clinically significant. One repeat evaluation of ECG, vital signs, and clinical laboratory tests will be permitted, at the discretion of the Investigator.
5. Subjects who test negative for hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (anti-HBc), anti-hepatitis C virus (HCV) antibodies, and anti-human immunodeficiency virus (HIV) 1 and 2 antibodies at Screening.
6. Subjects who test negative for SARS-Cov-2 infection, based on a reverse transcriptase polymerase chain reaction (RT-PCR) test and serological test for SARS-COV-2 IgM and/or IgG antibodies at Screening.
7. Female subjects are eligible to participate if not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

   1. Is not a woman of childbearing potential (WOCBP), defined as:

      Surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, as confirmed by review of the subject's medical records, medical examination, or medical history interview), or Postmenopausal (defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone [FSH] level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy [HRT]. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient). Female subjects on HRT and whose menopausal status is in doubt will be required to use 1 of the non estrogen hormonal highly effective contraception methods from Day 1 until at least 6 months after the second dose of IP if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.
   2. Is a WOCBP who agrees to use a highly effective method of contraception consistently and correctly from Day 1 until at least 6 months after the second dose of IP.
8. Nonsterilized male subjects with female partners of childbearing potential are eligible to participate if they agree to ONE of the following from Day 1 until at least 6 months after the second dose of IP and refrain from donating sperm during this period:

   1. Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.
   2. Agree to use a male condom and have their partner use of a contraceptive method with a failure rate of <1% per year when having penile-vaginal intercourse with a WOCBP who is not currently pregnant.
   3. Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration.

Exclusion Criteria:

* Subjects are excluded from the study if ANY of the following criteria apply at any time starting from Screening up to Day 1 prior to IP administration:

  1. History of clinically significant and uncontrolled hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurologic disease in the opinion of the Investigator within 12 months prior to Screening.
  2. Individuals with behavioral or cognitive impairment in the opinion of the Investigator.
  3. Individuals with any progressive or severe neurologic disorder, seizure disorder, or history of Guillain-Barré syndrome.
  4. Individuals with known or suspected impairment of the immune system, such as:

     1. Use of systemic (oral or parenteral) corticosteroids for ≥14 consecutive days within 60 days prior to Day 1. Use of inhaled, intranasal, or topical corticosteroids is allowed. NOTE: Systemic (oral or parenteral) corticosteroids are also prohibited for 3 weeks after the second dose of the IP.
     2. Receipt of cancer chemotherapy within 5 years prior to Day 1.
     3. Receipt of immunostimulants or immunosuppressants within 60 days prior to Day 1.
     4. Known HIV or acquired immune deficiency syndrome.
     5. Subjects with active or prior documented autoimmune disorder (such as potential immune mediated diseases [pIMDs]).
     6. Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Day 1 or planned during the full length of the study.
     7. Being treated for tuberculosis.
  5. History of allergic disease or reactions associated with previous vaccinations or likely to be exacerbated by any component of the IP.
  6. Individuals who have had a previous confirmed or suspected illness caused by SARS-CoV-1, SARS-CoV-2, or MERS-CoV.
  7. Individuals who have had a malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder within the past 5 years from the first dose of the IP (Day 1).
  8. History of urticaria within 1 year prior to Screening.
  9. History of hereditary angioneurotic edema or acquired angioneurotic edema.
  10. History of asplenia or functional asplenia.
  11. History of platelet disorder or other bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the Investigator, contraindicate intramuscular injection.
  12. Current febrile illness or body temperature ≥38.0°C or other moderate to severe illness within 24 hours of IP administration on Day 1. This condition is considered to be temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met.
  13. Any current active infections, including localized infections, or any recent history (within 1 week prior to IP administration) of active infections or cough; or a history of recurrent or chronic infections (>3 infections/year).
  14. Individuals with a history of drug or alcohol abuse (with an average intake exceeding 10 drinks/week for women and 15 drinks/week for men: 1 drink = 360 mL of beer, 150 mL of wine, or 45 mL of spirits) or drug addiction (including soft drugs like cannabis products) within the past 2 years.
  15. Current heavy smoker, defined as smoking ≥20 cigarettes/day (1 pack or equivalent), or a former heavy smoker who was an active smoker within the past 1 year prior to Screening.
  16. Individuals who faint at the sight of blood or needles.
  17. Participation in another interventional clinical study (including a bioequivalence study) with an investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of the IP.
  18. Individuals who have received any prior investigational or approved vaccine against a coronavirus, including but not limited to SARS-CoV-1, SARS-CoV-2, and MERS-CoV.
  19. Individuals who have received any other licensed vaccines within 14 days (for inactivated vaccines) or 30 days (for live or attenuated vaccines) prior to enrollment in this study, or those who are planning to receive any vaccine within 30 days before the first dose of IP or during the study, with the exception of the seasonal influenza vaccine.
  20. Individuals must not have donated blood for 30 days prior to Day 1 and must agree to not donate blood for 6 months after Day 1 (receipt of first dose of the IP).
  21. Individuals with any condition that, in the opinion of the Investigator, would interfere with the study objectives or pose additional subject risk.
  22. Any persons who are:

      1. An employee of the study site, Investigator, contract research organization (CRO) or Sponsor.
      2. A first-degree relative of an employee of the study site, the Investigator, CRO, or the Sponsor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with solicited local and systemic adverse events | up to 7 days after each dose
  Incidence of solicited local and systemic adverse events up to 7 days after each dose
Number of Participants with unsolicited adverse events after each dose | up to 30 days after the second dose
  Incidence of unsolicited adverse events after each dose up to 30 days after the second dose
Number of Participants with serious adverse events | up to 30 days after the second dose
  Incidence of serious adverse events up to 30 days after the second dose
Number of Participants with changes in clinical laboratory tests from baseline | up to 7 days after each dose
  Changes in clinical laboratory tests from baseline up to 7 days after each dose
Number of Participants with changes in vital signs from baseline | up to 30 days after the second dose
  Changes in vital signs from baseline up to 30 days after the second dose

SECONDARY OUTCOMES:
Number of Participants with adverse events,serious adverse events, and adverse events of special interest | up to 12 months after the second dose
  Incidence of adverse events,serious adverse events, and adverse events of special interest up to 12 months after the second dose
Number of Participants with changes in vital signs from baseline | up to 12 months after the second dose
  Changes in clinical laboratory tests and vital signs from baseline up to 12 months after the second dose
Geometric mean titers(GMT) | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  specific IgG binding antibodies against SARS-CoV-2
Seroconversion rates | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  specific IgG binding antibodies against SARS-CoV-2
Geometric mean fold increase | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  specific IgG binding antibodies against SARS-CoV-2
IFN-γ | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  Positivity rate of IFN-γ measured by ELISpot
Geometric mean titers(GMT) | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  specific IgG neutralizing antibodies against SARS-CoV-2
Seroconversion rates | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  specific IgG neutralizing antibodies against SARS-CoV-2
Geometric mean fold increase | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  specific IgG neutralizing antibodies against SARS-CoV-2
Levels of other T cell biomarkers | first dose day 21, second dose day 14, , day 30, day 90, day 180 and day 360
  CD4+/CD8+ counts, IL-4, IL-5, and IL-17

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wynne C, Balgos A, Li J, Hamilton P, Tirador L, Jaen AM, Mo C, Yue Z, Ma Y, Wang Q, Wen R, Yao Z, Yu J, Yao W, Zhang J, Zheng H, Hong K, Zhu F, Liu Y. Safety and Immunogenicity of a Recombinant Two-Component SARS-CoV-2 Protein Vaccine: Randomized, Double-Blind, Placebo-Controlled Phase I and Phase II Studies. Infect Dis Ther. 2024 Jan;13(1):57-78. doi: 10.1007/s40121-023-00896-w. Epub 2023 Dec 16. PMID 38103161